CLINICAL TRIAL: NCT01301027
Title: Effects of Pioglitazone on Adiponectin and Inflammatory Markers in Overweight or Obese Hemodialysis Patients: A Double-Blinded Randomized Controlled Trial
Brief Title: Effect of Adipokines in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Srinvasan Beddhu, MD, Associate Professor of Medicine, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB_00028427; R01DK078112 (NIH)
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Results first posted 2016-10-03 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-08

CONDITIONS: End Stage Renal Disease
Keywords: End stage renal disease; Hemodialysis; Pioglitazone; Adipokines
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone (Active Comparator): 15 mg/day pioglitazone for 2 weeks, then 30 mg/day for remaining 24 weeks
  Interventions: Drug: Pioglitazone
- Placebo (Placebo Comparator): 1 placebo pill a day matching the pioglitazone treatment for 26 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — 15mg/day pioglitazone for 2 weeks, then 30mg/day pioglitazone for the remaining 24 weeks
  Other Names: Actos
  Arms: Pioglitazone
Drug: Placebo — 1 pill a day for 26 weeks
  Arms: Placebo

SUMMARY:
This is a double blinded randomized clinical trial of pioglitazone vs. placebo in overweight or obese, diabetic and non-diabetic hemodialysis patients. This study will examine whether pioglitazone modulates adipokine production by adipose tissue in hemodialysis patients and whether these changes result in reduction of inflammation, insulin resistance and oxidative stress and increase in muscle mass.

In addition, this study will also examine the associations of adiposity with adipokines and the metabolic milieu in hemodialysis patients to better understand the biology of adipocytes in uremic milieu.

DETAILED DESCRIPTION:
Randomization:

100 overweight or obese patients will be randomly allocated to oral pioglitazone 15 mg/d or placebo for two weeks by blocks of five using a random number generator and monitored for adverse events including hypoglycemia. If they tolerate the 15 mg pioglitazone or matching placebo for two weeks, participants will be assigned to 30 mg of pioglitazone or matching placebo for 24 more weeks. Those who received 15 mg of pioglitazone will receive 30 mg of pioglitazone for the next 24 weeks. Those who received placebo for initial 2 weeks will receive another placebo that matches the 30 mg pioglitazone pill for 24 weeks.

Baseline:

Participants will have fasting blood drawn for adipokines: Tumor Necrosis Factor-alpha (TNF-alpha), Interleukin-6 (IL-6), high sensitivity C-Reactive Protein (hsCRP), high molecular weight Adiponectin (HMW-A), and leptin. All patients will undergo MRI scans on the mid-week non-dialysis day. Twenty each of overweight/obese patients randomized to pioglitazone or placebo will also undergo subcutaneous fat biopsy on the mid-week non-dialysis day.

Study Period:

Participants will return to the dialysis unit at weeks 2, 4, 6, 10, 14, 18, 22, and 26. During these visits, clinical assessments will be conducted including review of blood sugars, jaundice, weight gain, and visual symptoms. Study treatment compliance will be assessed and details of adverse events experienced, particularly hospitalizations and emergency department visits will be collected. Fasting blood draws for primary and secondary outcomes will be collected on visit weeks 10 and 26.

ELIGIBILITY:
Inclusion Criteria:

* Overweight (Body Mass Index ≥ 25 kilograms per meter squared (kg/m2))
* Adult (18 years or older)
* Chronic hemodialysis patient
* Diabetic (type 2) or insulin resistant

Exclusion Criteria:

* <18 years old
* No insulin resistance
* Active liver disease
* Class III or IV New York Heart Association heart failure
* Macular edema or hard exudates near macula on fundoscopy
* Current active malignancy (excluding squamous and basal cell skin cancers)
* Active AIDS
* Chronic lung disease requiring supplemental oxygen therapy
* Enrolled in interventional trials using drugs or devices
* Bone break of long bones, vertebrae, or hips in the past three years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2008-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srinivasan Beddhu, M.D., Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - University of Colorado, Denver, Colorado
  - University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pioglitazone | Placebo
Started | 48 | 47
Completed | 40 | 37
Not Completed | 8 | 10
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Fracture | 1 | 3
Not completed — Transplant | 0 | 2
Not completed — Volume Overload | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone | Placebo | Total
Number analyzed (Participants) | 48 | 47 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.17 (12.01) | 57.45 (14.12) | 58.32 (13.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 35 | 34 | 69
Body Mass Index [Mean (Standard Deviation); unit: kilograms per meter squared] | 32.3 (6.6) | 32.9 (7.5) | 32.6 (7.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in High Molecular Weight Adiponectin (HMW-A) Concentration in Plasma From Baseline to 6 Months
Description: The percent difference in HMW-A concentration geometric mean values from baseline to 6 months was calculated for each arm
Time Frame: Baseline and 6 months
Population: 1 participant in the Pioglitazone group and 2 participants in the Placebo group had blood samples collected after the 10 week visit prior to their withdrawal. They did not complete the study, but their results were included in the 6-month analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: percent difference in geometric mean
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 41 | 39
percent difference in geometric mean | 38.3 [4.9 to 82.2] | -3.4 [-27.0 to 27.8]
Statistical Analysis 1: Comparison: Pioglitazone vs Placebo; Test type: Superiority or Other; p = 0.047, t-test, 2 sided

2. Primary Outcome: Change in High Sensitivity C-Reactive Protein (hsCRP) Concentration in Plasma From Baseline to 6 Months
Description: The percent difference in hsCRP concentration geometric mean values from baseline to 6 months was calculated for each arm
Time Frame: Baseline and 6 months
Population: 1 participant in the Pioglitazone group and 2 participants in the Placebo group had blood samples collected after the 10 week visit and prior to their withdrawal. They did not complete the study, but their results were included in the 6-month analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: percent difference in geometric mean
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 41 | 39
percent difference in geometric mean | -29.0 [-44.7 to -8.8] | -1.8 [-23.8 to 26.5]
Statistical Analysis 1: Comparison: Pioglitazone vs Placebo; Test type: Superiority or Other; p = 0.059, t-test, 2 sided

3. Secondary Outcome: Change in Tumor Necrosis Factor-α (TNF-α) Concentration in Plasma From Baseline to 6 Months
Description: The percent difference in TNF-α concentration geometric mean values from baseline to 6 months was calculated for each arm
Time Frame: Baseline and 6 months
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: percent difference in geometric mean
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 41 | 39
percent difference in geometric mean | 44.9 [32.9 to 58.1] | 39.1 [27.3 to 51.9]
Statistical Analysis 1: Comparison: Pioglitazone vs Placebo; Test type: Superiority or Other; p = 0.508, t-test, 2 sided

4. Secondary Outcome: Change in Interleukin-6 (IL-6) Concentration in Plasma From Baseline to 6 Months
Description: The percent difference in IL-6 concentration geometric mean values from baseline to 6 months was calculated for each arm
Time Frame: Baseline and 6 months
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: percent difference in geometric mean
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 41 | 39
percent difference in geometric mean | -12.3 [-29.7 to 9.6] | -12.5 [-30.1 to 9.5]
Statistical Analysis 1: Comparison: Pioglitazone vs Placebo; Test type: Superiority or Other; p = 0.984, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 26 Weeks
Description: Details of adverse events experienced, particularly hospitalizations and emergency department visits obtained at each scheduled follow-up visit through Week 26
Arm/Group | Pioglitazone | Placebo
Serious Adverse Events (participants affected / at risk) | 11/48 | 10/47
Other Adverse Events (participants affected / at risk) | 16/48 | 6/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=48) | Placebo (N=47)
Cardiac General - Volume Overload (Cardiac disorders) | 0 (0) | 2 (2)
Death (General disorders) | 1 (1) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Flu-like Syndrome (General disorders) | 1 (1) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Colon Cancer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhage - Lower GI NOS (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Infection - Blood (Bacteremia) (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain NOS (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chext/Thorax Pain NOS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pancreatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Fistula failure (Vascular disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=48) | Placebo (N=47)
Cardiac General - Volume Overload (Cardiac disorders) | 4 (4) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 4 (5) | 1 (1)
Dizziness (Nervous system disorders) | 3 (5) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (9) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (9) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No